CLINICAL TRIAL: NCT04530331
Title: Work-Site Nutrition Education and Metabolic Syndrome Factors
Brief Title: Job-Site Diet Education on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Principal Investigator, Hsien-Cheng Chang, Director, Lotung Poh-Ai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lotung Poh-Ai Hospital
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Metabolic Syndrome; Health Education; Workplace
MeSH Terms: conditions — Metabolic Syndrome; Health Education | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Providing nutrition education.
  Interventions: Behavioral: Nutrition education
- Control group (No Intervention): Without any intervention.

INTERVENTIONS:
Behavioral: Nutrition education — Dietitians visited the worksites of the intervention group once a week to deliver a nutrition education session and provide dietary advice for each participant.
  Arms: Intervention group

SUMMARY:
This study conducted an 8-week workplace nutrition education intervention to examine the effects of the intervention on metabolic syndrome factors associated with employees. A historical intervention was designed to recruit adults with a body mass index level of >22 and without any endocrine disorder from a community in Yilan, Taiwan. The intervention group was recruited between 2010 and 2012 and received an 8-week intervention, during which dietitians delivered a nutrition education session and a one-on-one dietary guidance session on a weekly basis. The age- and sex-matched control group (n = 34) was recruited between 2014 and 2015 to analyze the metabolic syndrome variables. The metabolic syndrome variables included blood pressure, blood sugar, serum lipid profile, and waist circumference.

DETAILED DESCRIPTION:
Content of classes Week1 Things that you must know during the weight reduction study period Week2 Daily individual calorie requirement: what are the main food groups? Week3 How to record the daily diet after the weight reduction program Week4 Food serving size and replacement Week5 The principles of eating out Week6 Physical activity advice (delivered with health education flyers to the participants)

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* BMI of ≥ 22

Exclusion Criteria:

* History of critical illness
* Having been diagnosed with at least one endocrine disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2010-03-08 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
BMI | After 8 week intervention
  To evaluate the effect of nutrition education on the reduction of BMI (body mass index).
Waist circumference | After 8 week intervention
  One of the metabolic syndrome factors.
Systolic blood pressure | After 8 week intervention
  One of the metabolic syndrome factors.
Diastolic blood pressure | After 8 week intervention
  One of the metabolic syndrome factors.
Fasting blood sugar | After 8 week intervention
  One of the metabolic syndrome factors.
Serum triglyceride | After 8 week intervention
  One of the metabolic syndrome factors.
Serum high density lipoprotein cholesterol | After 8 week intervention
  One of the metabolic syndrome factors.